CLINICAL TRIAL: NCT04693767
Title: Investigation of Clot in Ischemic Stroke and Hematoma Evacuation
Acronym: INSIGHT
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 15131
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke; Intracranial Hematoma
MeSH Terms: conditions — Ischemic Stroke | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Clot and blood specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Patients with ischemic stroke
  Interventions: Device: Mechanical thrombectomy
- Patients with intracranial hematoma
  Interventions: Other: Minimally invasive surgery

INTERVENTIONS:
Device: Mechanical thrombectomy — 1. Clot specimen collection
  2. Extracranial blood collection
  Groups: Patients with ischemic stroke
Other: Minimally invasive surgery — 1. Clot specimen collection
  2. Arterial blood collection
  Groups: Patients with intracranial hematoma

SUMMARY:
The aim of the study is to collect and analyze specimen from ischemic stroke patients undergoing thrombectomy procedures and from patients undergoing minimally invasive surgery for intracranial hematoma evacuation.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 Years of Age
* Frontline treatment with: Penumbra System for ischemic stroke patients eligible for mechanical thrombectomy or Artemis Neuro Evacuation device for intracranial hematoma evacuation in patients eligible for minimally invasive surgery (MIS)
* Extracted thrombus/embolus
* Informed consent is obtained from either the patient or legally authorized representative (LAR)

Exclusion Criteria:

* Pregnancy or positive pregnancy test according to site routine practice (only required for women of child bearing potential; serum or urine acceptable)
* Currently participating in an investigational drug or device clinical trial that may confound the ability to capture clot and/or influence clot composition. Patients in observational, natural history, and/or epidemiological studies not involving intervention are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing either ischemic stroke thrombectomy procedures or minimally invasive interventions for intracranial hematoma evacuation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner University Medical Center - Phoenix, Phoenix, Arizona
  - Christiana Care, Newark, Delaware
  - George Washington University, Washington D.C., District of Columbia
  - Baptist Medical Center, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Norton Neuroscience Institute, Louisville, Kentucky
  - MaineHealth, Portland, Maine
  - Adventist Healthcare Shady Grove Medical Center, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Metro Health, Wyoming, Michigan
  - St. Dominic Jackson Memorial Hospital, Jackson, Mississippi
  - SSM St. Clare Healthcare, Fenton, Missouri
  - Mount Sinai, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Westchester Medical Center, Valhalla, New York
  - Miami Valley Hospital, Dayton, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Memorial / Prisma Health, Greenville, South Carolina
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - Methodist University, Memphis, Tennessee
  - University of Texas Health Center, Memorial Hermann Medical Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Health Services, Swedish Cherry Hill, Seattle, Washington
  - Tacoma General Hosptial, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Ischemic Stroke: Mechanical thrombectomy
- Patients With Intracranial Hematoma: Minimally invasive surgery
Period: Overall Study
Arm/Group | Patients With Ischemic Stroke | Patients With Intracranial Hematoma
Started | 388 | 12
Completed | 388 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Ischemic Stroke: Mechanical thrombectomy: 1) Clot specimen collection 2) Extracranial blood collection
- Patients With Intracranial Hematoma: Minimally invasive surgery: 1) Clot specimen collection 2) Arterial blood collection
- Total: Total of all reporting groups
Arm/Group | Patients With Ischemic Stroke | Patients With Intracranial Hematoma | Total
Number analyzed (Participants) | 388 | 12 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (14.85) | 61.9 (11.65) | 68.9 (14.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 3 | 206
  Male | 185 | 9 | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 13
  Not Hispanic or Latino | 360 | 7 | 367
  Unknown or Not Reported | 19 | 1 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 73 | 2 | 75
  White | 276 | 3 | 279
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 31 | 5 | 36

OUTCOME MEASURES:

1. Primary Outcome: Clot Specimen Histology
Description: Numbers of clot specimen for histology analysis
Time Frame: Clot specimen obtained during procedure
Population: Total of 388 participants in Ischemic Stroke Cohort and 12 participants in Intracranial Hematoma Cohort.
Measure: Number; unit: Count of specimen
Groups:
- Patients With Ischemic Stroke; Patients With Intracranial Hematoma: Clot Histology
Arm/Group | Patients With Ischemic Stroke | Patients With Intracranial Hematoma
Number analyzed (Participants) | 388 | 12
Count of specimen | 373 | 12

2. Primary Outcome: Blood and Clot Specimen Transcriptomics
Description: Numbers of blood and clot for RNA sequency. Only includes successful sample number that was processed.
Time Frame: Blood and clot specimen obtained during procedure
Population: Total of 388 participants in Ischemic Stroke Cohort and 12 participants in Intracranial Hematoma Cohort.
Measure: Number; unit: Count of specimen
Groups:
- Patients With Ischemic Stroke; Patients With Intracranial Hematoma: Clot RNA Analysis and Blood RNA Analysis
Arm/Group | Patients With Ischemic Stroke | Patients With Intracranial Hematoma
Number analyzed (Participants) | 388 | 12
Count of specimen
  Clot RNA Analyzed | 341 | 9
  Blood RNA Analyzed | 365 | 12

3. Primary Outcome: Blood and Clot Specimen Proteomics
Description: Numbers of blood and clot specimen for proteomic analysis
Time Frame: Blood and clot specimen obtained during procedure
Population: Total of 388 participants in Ischemic Stroke Cohort and 12 participants in Intracranial Hematoma Cohort.
Measure: Number; unit: Count of specimen
Groups:
- Patients With Ischemic Stroke; Patients With Intracranial Hematoma: Clot Protein Analysis and Blood Protein Analysis
Arm/Group | Patients With Ischemic Stroke | Patients With Intracranial Hematoma
Number analyzed (Participants) | 388 | 12
Count of specimen
  Clot Protein Analysis | 351 | 12
  Blood Protein Analysis | 366 | 12

4. Primary Outcome: Blood and Clot Specimen Genomics
Description: Numbers of blood and clot specimen for single nucleotide polymorphisms (SNPs). Only includes successful sample number that was processed.
Time Frame: Blood and clot specimen obtained during procedure
Population: Total of 388 participants in Ischemic Stroke Cohort and 12 participants in Intracranial Hematoma Cohort.
Measure: Number; unit: Count of specimen
Groups:
- Patients With Ischemic Stroke; Patients With Intracranial Hematoma: SNP Analysis
Arm/Group | Patients With Ischemic Stroke | Patients With Intracranial Hematoma
Number analyzed (Participants) | 388 | 12
Count of specimen | 387 | 12

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 7 days post-procedure.
Description: Adverse Event (AE): any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in participants, whether anticipated or unanticipated. As was pre-specified in the study protocol, only participants with Ischemic Stroke, who were treated with a RED Reperfusion Catheter (N=165), were assessed for serious and other adverse events. The RED Reperfusion Catheter was not a treatment option for participants with Intracranial Hematoma.
Arm/Group | Patients With Ischemic Stroke | Patients With Intracranial Hematoma
All-Cause Mortality (participants affected / at risk) | 86/388 | 3/12
Serious Adverse Events (participants affected / at risk) | 38/165 | 0/0
Other Adverse Events (participants affected / at risk) | 11/165 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Ischemic Stroke (N=165) | Patients With Intracranial Hematoma (N=0)
Symptomatic ICH (Nervous system disorders) | 4 | NA
Acute Ischemic Stroke (Nervous system disorders) | 5 | NA
Hemorrhagic Stroke (Nervous system disorders) | 1 | NA
Progression of Index Stroke (Nervous system disorders) | 13 | NA
New or Worsening Neurological Deficit (Nervous system disorders) | 3 | NA
Pneumonia (Infections and infestations) | 5 | NA
Other (Investigations) | 7 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Ischemic Stroke (N=165) | Patients With Intracranial Hematoma (N=0)
Anemia (Blood and lymphatic system disorders) | 1 | NA
Progression of Index Stroke (Nervous system disorders) | 3 | NA
Asymptomatic ICH (Nervous system disorders) | 5 | NA
Asymptomatic Petechial Hemorrhage (Nervous system disorders) | 2 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04693767/Prot_SAP_000.pdf